CLINICAL TRIAL: NCT05437575
Title: Prehospital Analgesia INtervention Trial (PAIN)
Acronym: PAIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jason Sperry (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jason Sperry, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY22010164; HT9425-25-F-0041 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-05-24; First posted 2022-06-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Traumatic Injury
Keywords: Trauma; ketamine hydrochloride; fentanyl citrate; shock; pain
MeSH Terms: conditions — Wounds and Injuries; Shock; Pain | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine Hydrochloride (Experimental): 2 blinded doses 2.5mg/ml ketamine hydrochloride in separately sealed pre-filled syringes Subjects will be administered the first dose over approximately 2 minutes via slow IV push. Pain assessment following administration will be obtained and recorded every 15 minutes. Redosing may occur after approximately 15 minutes if the subject has a qualifying pain score, there are no contraindications to pain medication per local protocol, and no exclusion criteria have been met.
  Interventions: Drug: Ketamine Hydrochloride
- Fentanyl Citrate (Active Comparator): 2 blinded doses 10mcg/ml in separately sealed pre-filled syringes Subjects will be administered the first dose over approximately 2 minutes via slow IV push. Pain assessment following administration will be obtained and recorded every 15 minutes. Redosing may occur after approximately 15 minutes if the subject has a qualifying pain score, there are no contraindications to pain medication per local protocol, and no exclusion criteria have been met.
  Interventions: Drug: Fentanyl Citrate

INTERVENTIONS:
Drug: Ketamine Hydrochloride — ketamine hydrochloride 2.5mg/ml packaged in pre-filled syringe
  Arms: Ketamine Hydrochloride
Drug: Fentanyl Citrate — fentanyl citrate 10mcg/ml packaged in pre-filled syringe
  Arms: Fentanyl Citrate

SUMMARY:
The Prehospital Analgesia INtervention trial (PAIN) is a proposed 4 year (3-year enrollment) multicenter, prehospital, randomized, double-blind, clinical trial that will enroll approximately 994 patients at select LITES Network sites. The objective is to perform a prospective, interventional, randomized trial among prehospital trauma patients with compensated shock (SI≥0.9 or HR ≥115) and an indication for pain management, comparing patient centered outcomes following prehospital administration of ketamine hydrochloride versus fentanyl citrate.

ELIGIBILITY:
Inclusion Criteria:

* Transport after injury to a participating PAIN Trauma center
* 2. Patient with compensated shock as defined by Shock Index (SI) ≥0.9 or Heart Rate (HR) ≥115.
* Intravenous pain medication indicated (CPOT≥2, NRS≥5) prior to arrival at the trauma center

Exclusion Criteria:

* No IV access
* Age <18 years
* Females <50 years of age
* SBP>180 mmHg at time of enrollment
* Advanced airway management prior to first dose administration
* Known allergy to fentanyl citrate or ketamine hydrochloride
* Known prisoner
* Objection to study voiced by subject or family member at scene
* Pain treatment contraindicated by local protocol
* Wearing a "NO PAIN STUDY" bracelet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 994 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
24-hour mortality | trauma bay arrival through 24 hours
  All cause mortality within 24 hours from time of trauma bay arrival

SECONDARY OUTCOMES:
Hypoxia | from initial administration of PAIN prehospital analgesia through hospital arrival
  incidence of hypoxia in the prehospital environment
Hypotension | from initial administration of PAIN study prehospital analgesia through hospital arrival
  incidence of hypotension in the prehospital environment
Need for airway management | from initial administration of PAIN study prehospital analgesia through hospital arrival
  need for airway management in the prehospital environment
Prehospital pain assessment following analgesia | from initial administration of PAIN study prehospital analgesia through hospital arrival
  prehospital pain assessment using Numeric Rating Scale (NRS)/Critical Care Pain Observational Tool (CPOT) scores. For Numeric Rating Scale, the patient rates their pain on a scale of 0 to 10 where 0 is no pain and 10 is the worst pain. The Critical Care Pain Observation Tool is used for patients who are intubated and cannot verbalize a pain score. Medical staff will observe the patient's behavior and score the patient's pain on a scale of 0 to 10, where 0 is no pain and 10 is the worst pain.
Trauma bay arrival pain score | score assessed at time of arrival to trauma bay
  pain assessment using Numeric Rating Scale (NRS)/Critical Care Pain Observation Tool (CPOT) score. For Numeric Rating Scale, patients rate their pain on a scale of 0 to 10 where 0 is no pain and 10 is the worst pain. The Critical Care Pain Observation Tool is used for patients who are intubated and cannot verbalize a pain score. A nurse will observe behavior and score the patient's pain on a scale of 0 to 10 where 0 is no pain and 10 is the worst pain.
Number of analgesic doses necessary to reduce pain level to <5 NRS or CPOT less than 2 | from initial administration of PAIN study prehospital analgesia through hospital arrival
  Number of analgesic doses necessary to reduce pain level to <5 on Numeric Rating Scale or less than 2 on Critical Care Pain Observation Tool. For Numeric Rating Scale, the patient rates their pain on a scale of 0 to 10 where 0 is no pain and 10 is the worst pain. The Critical Care Pain Observation Tool is used for patients who are intubated and cannot verbalize a pain score. A nurse will observe behavior and score the patient's pain on a scale of 0 to 10 where 0 is no pain and 10 is the worst pain.
24 hour opioid use | from initial administration of PAIN study prehospital analgesia through 24 hours
  total 24 hour opioid use
Incidence of prehospital adverse events | from initial administration of PAIN study prehospital analgesia through hospital arrival
  Incidence of adverse events of allergic reaction, emergence, laryngospasm, dysphoria, pruritus, and nausea
Survival to hospital discharge | administration of PAIN study prehospital analgesia through hospital discharge or death up to 30 days
  survival to hospital discharge
Ventilator free days | from administration of PAIN study prehospital analgesia through hospital discharge or death up to 30 days
  ventilator free days. Ventilator days are defined as number of days recorded to the first decimal spent on a mechanical ventilator subtracted from 30
Intensive Care Unit free days | from administration of PAIN study prehospital analgesia through hospital discharge or death up to 30 days
  number of days recorded to the first decimal spent admitted to the Intensive Care Unit subtracted rom 30
Long term opioid use | 3 months (+/- 1 month) and 6 months (+/- 1 month) following trauma admission
  long term opioid use assessed at 3 and 6 months. Patients who consent to further participation will be contacted to determine if they continued to use opioids (yes/no) at 3 and 6 months following trauma admission
Hospital length of stay | from time of hospital admission to discharge
  number of days recorded to the first decimal from hospital admission to discharge up to 30 days
Baseline Pain/Anxiety/PTSD screening | 0 hours to 2 weeks from time of hospital admission
  A subset of patients who consent to further participation will be assessed for Anxiety/PTSD using the Four-Item Patient Health Questionnaire (PHQ-4) for anxiety and depression, a two item pain severity scale (0=no pain to 10=worst pain), and the Injured Trauma Survivor Screen (ITSS)
Long term (6 month) outcome | 6 months +/- 1 month following trauma admission
  A subset of patients who consent to further participation will be assessed for anxiety/depression/PTSD symptoms using the following tools: Generalized Anxiety Disorder (GAD-7), 8 item Patient Health Questionnaire (PHQ-8), and 8 item PTSD checklist (PCL-5)
Long Term Pain Assessment | At 3 and 6 months (+/- 1 month) after hospital arrival
  A subset of patients who consent to further participation will be assessed for long term pain using a modified Brief Pain Inventory (numerical scale rating 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sperry, MD, Principal Investigator — University of Pittsburgh
Locations (10):
- United States (10):
  - University of California, San Diego, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - Cooper University Health Care, Camden, New Jersey
  - Atrium Health and Carolinas Medical Center, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Allegheny Health Network (AHN) Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Guthrie Robert Packer Hospital, Sayre, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with the funding agency as well as other researchers upon request to the Principal Investigator
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after publication of the primary manuscript
Access Criteria: Requests for data will be submitted in writing and reviewed by the Principal Investigator.